CLINICAL TRIAL: NCT05032833
Title: A Double-Blind, Randomized, Phase 1, First-in-Human, Single Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetic Profile of Intranasal 5-Methoxy-N,N-dimethyltryptamine (5-MeO-DMT) in Healthy Subjects
Brief Title: Single Ascending Dose Study With 5-MeO-DMT in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beckley Psytech Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BPL-5MEO-101
Record Dates: First submitted 2021-08-24; First posted 2021-09-02 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Pharmacokinetics in Healthy Adults
MeSH Terms: interventions — Methoxydimethyltryptamines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5-MeO-DMT arm (Experimental)
  Interventions: Drug: 5-MeO-DMT
- Placebo arm (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 5-MeO-DMT — A single dose of 5-MeO-DMT will be administered intranasally
  Arms: 5-MeO-DMT arm
Other: Placebo — A single dose of placebo will be administered intranasally
  Arms: Placebo arm

SUMMARY:
The study will evaluate safety, tolerability and PK profile of 5-MeO-DMT in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy based on medical records and study specific assessments

Exclusion Criteria:

* Presence or history of severe adverse reaction to any drug or drug excipient

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with treatment emergent AEs (TEAES) | From screening through to the follow up visit, up to 65 days

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) | Day 1 (dosing day) and Day 2
Time to reach Cmax (tmax) | Day 1 (dosing day) and Day 2
Area under the plasma concentration- time curve | Day 1 (dosing day) and Day 2

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Due to the UK GDPR, individual participant data will not be shared publicly. Group data will be presented in publication after study completion